CLINICAL TRIAL: NCT02232594
Title: Postmarketing Surveillance Study (as Per § 67 (6) AMG [German Drug Law]) of Berodual® Metered-dose Inhaler in Chronic Obstructive Respiratory Tract Disease
Brief Title: Postmarketing Surveillance Study of Berodual® Metered-dose Inhaler in Chronic Obstructive Respiratory Tract Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 215.1358
Record Dates: First submitted 2014-09-04; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fenoterol, ipratropium drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- chronic obstructive respiratory tract disease patients
  Interventions: Drug: Berodual®

INTERVENTIONS:
Drug: Berodual®

SUMMARY:
The aim of this postmarketing surveillance is to obtain further information about the tolerability and efficacy of Berodual® metered-dose inhaler in the treatment of chronic obstructive respiratory tract disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex over 40 years with the symptoms of a chronic obstructive airways disease
* Only patients which have not been treated with Berodual® within the last year should be included

Exclusion Criteria:

* Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Berodual® metered-dose inhaler

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive respiratory tract disease recruited at general physicians and internists
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2000-01; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Overall severity of the clinical picture rated on a 4- point scale | after 3 and 6 weeks

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 4-point scale | after 3 and 6 weeks
Assessment of efficacy by patient on a 4-point scale | after 3 and 6 weeks
Assessment of tolerability by investigator on a 4-point scale | after 3 and 6 weeks
Assessment of tolerability by patient on a 4-point scale | after 3 and 6 weeks
Number of patients with adverse drug reactions | up to 6 weeks